CLINICAL TRIAL: NCT03197402
Title: Efficacy of a High Quality Protein Leucine-enriched Nutraceutical in Attenuating Inactivity- and Hypo-energetic Diet-induced Muscle Loss in Older Women
Brief Title: Leucine-enriched Nutraceutical and Attenuating Muscle Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3390
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Muscle Loss
Keywords: Leucine; Protein; Supplementation
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: parallel group design (with repeated measurements within each group)
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator group (Active Comparator): Milk protein gel delivery system supplementation
  Interventions: Dietary Supplement: Milk protein gel delivery system
- Leucine-enriched protein group (Experimental): Leucine-enriched protein gel delivery system supplementation
  Interventions: Dietary Supplement: Leucine-enriched protein gel delivery system

INTERVENTIONS:
Dietary Supplement: Leucine-enriched protein gel delivery system — Leucine enriched
  Arms: Leucine-enriched protein group
Dietary Supplement: Milk protein gel delivery system — Non-leucine enriched
  Arms: Comparator group

SUMMARY:
This leucine-enriched protein gummy (as a gummy bar/slab) will be studied to address age-related loss of muscle mass and strength/function in older persons. The product is small volume (approximately 35 g per serve) and low energy (approximately 100 kcal per serve). It is easy to chew and swallow with the consistency of a firm Jello. In addition, it contains an effective dose of leucine in a high-quality protein matrix consisting of milk proteins. Understanding the efficacy of this product on changes in levels of blood amino acids and the molecular signaling required to enhance muscle growth will provide helpful insight for the suggestion of supplemental use.

DETAILED DESCRIPTION:
General experimental design:

Pre-testing will require participants to become familiarized with performing maximal voluntary isometric contractions, as well as touring the laboratory facilities. Participants will be asked to complete dietary records for three days to determine habitual caloric intake. The experimental trial will be conducted in three phases. A baseline run-in phase (Phase 1) during which participants will consume a diet matching their estimated energy requirement to put them in a weight-stable phase. Energy requirements will be estimated using the Harris Benedict equation using an appropriate physical activity factor based on interview responses to a standard activity questionnaire. Participants will then be assigned to either the comparator group (n=10) or leucine-enriched protein food group (n=10). For the subsequent 10d (Phase 2), participants will undergo a period of step reduction (< 1000 steps.d-1) whilst in a 500 kcal.d-1 deficit that will be adjusted for the reduced physical activity due to the step reduction. The reason for inducing an energy deficit is to mimic a situation where older individuals will be both physically inactive and 'undernourished', such as during home-bound periods of sickness or while in hospital. After completing Phase 2, participants will then return to their normal step count (from measured habitual steps pre-intervention) under energy balanced conditions for 10d that will serve as a recovery phase, Phase 3. We will complete assessments of body composition, leg lean mass, maximal voluntary isometric strength, measures of physical performance, and rate of force development will be made. Skeletal muscle biopsies will be obtained for biochemical analysis. At these time points, maximal voluntary isometric force, maximal leg press strength, a battery of physical performance measures and body composition will once again be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Females between 70 and 75 years of age (a narrow age range improved homogeneity of the sample for this proof-of-concept trial) with a body mass index (BMI) between 27 and 35, and muscle mass 1 standard deviation below that of sex- and ethnicity-matched 30 year olds (note: this has been called 'stage 1 sarcopenia' or 'pre-sarcopenia') will be recruited. In addition, participants will be non-smokers and generally healthy per responses to a standard health screening questionnaire.

Exclusion Criteria:

* Participants who have any one of the following conditions will be excluded:

  * diabetes mellitus
  * cardiovascular disease
  * renal disease
  * gastrointestinal disease
  * musculoskeletal injuries
  * hormone replacement therapy
  * significant weight loss in the 3-month period prior to the study
  * vegan diet
  * dairy protein allergy
  * use of medications known to interfere with muscle metabolism. For example, chronically taking any analgesic or anti-inflammatory drugs(s), prescription or non-prescription
  * a history of neuromuscular problems or muscle and/or bone wasting diseases
  * any acute or chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, insulin- or non-insulin dependent diabetes or other metabolic disorders-all ascertained through medical history screening questionnaires
  * use medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications)

Ages: 70 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline molecular signalling | Through study completion, an average of 1 year
  protein synthetic pathway

SECONDARY OUTCOMES:
Change from baseline lean body mass | Through study completion, an average of 1 year
  body composition

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario
  - Ivor Wynne Centre A103, McMaster University, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No
These data will not be shared with other researchers

REFERENCES:
- [Result] Sullivan DH, Sun S, Walls RC. Protein-energy undernutrition among elderly hospitalized patients: a prospective study. JAMA. 1999 Jun 2;281(21):2013-9. doi: 10.1001/jama.281.21.2013. PMID 10359390